CLINICAL TRIAL: NCT06307444
Title: Ultrasound-Guided Erectro Spinae Plane Block Versus Stellate Ganglion Block for Patients With Upper Limb Acute Herpes Zoster Pain: Randomized Controlled Study
Brief Title: Ultrasound-Guided Erectro Spinae Plane Block Versus Stellate Ganglion Block for Patients With Upper Limb Acute Herpes Zoster Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aliaa Muhammad Belal, Principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: stellate block and ESP block
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acute Herpes Zoster Pain Managment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- medical treatment only (No Intervention): All patients will receive oral medication for antiviral therapy (800mg of acyclovir 5 times daily) at the time of diagnosis and supportive treatments, including acetaminophen (1gm 3times daily), and gabapentin (starting at 100mg three times daily) to be incrementally up titrated over time as needed by 100 to 300 mg every 3 to 5 days, to as high a dosage as 1800 to 3600 mg/day in 3 or 4 divided doses
- Ultrasound-Guided Stellate Ganglion Block (Experimental): Ten milliliters of a local anesthetic solution (bupivacaine (0.25%)+ 8 mg dexamethasone) is injected until the fluid spreads along the paravertebral fascia to the stellate ganglion.
  Interventions: Procedure: Ultrasound-Guided Stellate Ganglion Block
- Group III T2 T3 (High Thorathic) ErectroSpinae Plan Block (Experimental): ocal anesthetic drugs(0.2-0.3ml/kg of bupivacaine 0.25% 8mg Dexamethazone) will be administered as standard in all patients aiming to distribute within the plane between the anterior fascia of the erector spinae muscle and the transverse process.
  Interventions: Procedure: T2 T3 (High Thorathic) ESP Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Stellate Ganglion Block — high frequency (6 to 13 MHz) linear transducer will be placed perpendicular to the tracheal axis at the cricoid cartilage and will be moved inferiorly until the superior aspect of the thyroid gland is visualized. Later, the transducer should be relocated laterally to visualize the anterior aspect of the Chassaignac's tubercle on []the C6 transverse process. The carotid artery, internal jugular vein, thyroid gland, trachea, Longus colli, and Longus capitis muscle, prevertebral fascia, the root of C6 spinal nerve, and transverse process of C6 can be identified. Color Doppler will be used to detect the position of the vessels. With an in-plane approach, 22 to 25 gauge echo-enhanced needle is placed beside the trachea with a lateral to medial direction.
  Arms: Ultrasound-Guided Stellate Ganglion Block
Procedure: T2 T3 (High Thorathic) ESP Block — We will count the laminae in the cephaled-to-caudal direction, starting from the C7 using the US to determine the exact vertebral level where the needle will be inserted. A linear high-frequency ultrasound probe will be used to perform the blocks. After the determination of the needle insertion site, the US probe was placed over the spinous processes of the vertebrae at the midline in the longitudinal plane. The US probe will then slid laterally from the spinous processes to visualize the transverse process. The needle will be advanced posterior-to-anteriorly, in the caudal to cephalic direction using the in-plane orientation within paraspinal muscles, targeting the transverse process. When the tip of the needle reaches and contact the transverse process, the local anesthetic drugs(0.2-0.3ml/kg(11) of bupivacaine 0.25% 8mg Dexamethazone) will be administered
  Arms: Group III T2 T3 (High Thorathic) ErectroSpinae Plan Block

SUMMARY:
Herpes zoster (HZ) is a painful, eruptive, viral condition results from reactivation of the latent varicella zoster virus after the primary infection. The selection of an effective analgesic method in the acute phase of herpes zoster can decrease the incidence of postherpetic neuralgia by reducing neural sensitization. The stellate ganglion is present in 80% of the general population and is composed of the inferior cervical ganglion and the first thoracic ganglion fusion. It lies anterior to the neck of the first rib and extends to the inferior aspect of the transverse process of C7. The erector spinae plane (ESP) block has been reported to provide diffuse and effective analgesia in the cervical, thoracic, and lumbar regions.

DETAILED DESCRIPTION:
Especially for elderly patients, when cell-mediated immunity wanes, common symptoms of HZ appear, primarily as pain in a dermatomal distribution with a burning, sharp pain sensation (paresthesia) and itching, in addition to development of a vesicular rash. The selection of an effective analgesic method in the acute phase of herpes zoster can decrease the incidence of postherpetic neuralgia by reducing neural sensitization. The sympathetic fibers for the head, neck, heart, and upper limbs arise from the first thoracic segments, ascend through the sympathetic chain, and synapse in the superior, middle, and inferior cervical ganglions. The stellate ganglion is present in 80% of the general population and is composed of the inferior cervical ganglion and the first thoracic ganglion fusion. It lies anterior to the neck of the first rib and extends to the inferior aspect of the transverse process of C7. The erector spinae plane (ESP) block has been reported to provide diffuse and effective analgesia in the cervical, thoracic, and lumbar regions.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 21 with upper limb herpetic eruption lasting shorter than a week along with moderate to severe pain who got adequate antiviral medications

Exclusion Criteria:

* We will exclude patients who refuse to participate, those who are taking anticoagulant medications, have secondary bacterial infections of the dermatome, those who have an allergy to local anesthetics or serious disease of the heart ( e.g. heart block), lung, kidneys and those who had a history of neck surgery, such as thyroid cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
reduction of a numeric rating scale (NRS) pain score | after the porcedure till 12 weak
  1. Pain intensity before block by NRS score (0-10)
  2. Pain intensity after block by NRS score (0-10) Pain intensity at 1,2,3,4, ,6,8,12 and24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa M Belal, MD, Principal Investigator — tanta univ
Locations (1):
- Tanta university faculty of medicine, Tanta, None Selected, Egypt